CLINICAL TRIAL: NCT04229121
Title: Clinical Sensitivity Verification Study of Circulating Tumor Cells Gene Mutation Detection From Advanced NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Director Head of Medical Oncology, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: CTC-FM
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Advanced NSCLC; Circulating Tumor Cells; Circulating Tumor DNA
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Driver gene mutation-positive: Screen the enrolled patients according to the admission criteria. The detection of lung cancer Polymerase Chain Reaction (PCR) panel kit in the hospital requires the use of tissue samples and the results show a Driver gene mutation positive.
  Interventions: Other: nonintervention
- Driver gene mutation-negative: Screen the enrolled patients according to the admission criteria. The detection of lung cancer Polymerase Chain Reaction (PCR) panel kit in the hospital requires the use of tissue samples and the results show a Driver gene mutation negative.
  Interventions: Other: nonintervention

INTERVENTIONS:
Other: nonintervention — nonintervention

SUMMARY:
Verify the Coincidence rate between Circulating tumor cells (CTCs) and tumor tissue or Circulating tumor DNA (ctDNA) of advanced NSCLC patients with Driver gene mutation

DETAILED DESCRIPTION:
1. Enrich CTCs from advanced Non-Small Cell Lung Cancer (NSCLC) patients with Driver gene mutation, and detect the Epidermal Growth Factor Receptor (EGFR) mutation, Anaplastic lymphoma kinase (ALK) fusion, ROS proto-oncogene receptor tyrosine kinase 1 (ROS1) fusion, RET proto-oncogene (RET) fusion and Mesenchymal-Epithelial Transition factor (MET) 14 exon skipping by Lung cancer Polymerase Chain Reaction (PCR) panel kit, and verify the mutation coincidence rate between CTCs and tumor tissue.
2. Enrich ctDNA from advanced NSCLC patients with Driver gene mutation, detect the EGFR mutation by PCR, and detect the ALK fusion, ROS1 fusion, RET fusion and MET 14 exon skipping by next generation sequencing (NGS), and compare the mutation coincidence rate between CTCs and ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, 18 years of age or older
2. Histologically or cytologically proven diagnosis of advanced NSCLC patients without any target therapy or chemotherapy
3. Able to get tumor tissue gene (EGFR/ALK/ROS1/RET/MET skipping) testing results by Lung cancer Polymerase Chain Reaction (PCR) panel kit carried out in hospital
4. Signed and dated informed consent

Exclusion Criteria:

1. Combine with other tumor type
2. The investigator judges the situation that may affect the clinical search process and results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologially or cytologically proven diagnosis of advanced NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Driver gene mutation frequency from CTCs of advanced NSCLC patients | 6 months
  Analyze the driver gene mutation frequency in CTCs from advanced NSCLC patients with tumor tissue driver gene mutation
The gene mutation coincidence rate between CTCs and tumor tissue sample | 6 months
  Comparison the gene mutation coincidence rate between CTCs and tumor tissue sample

SECONDARY OUTCOMES:
Driver gene mutation frequency from ctDNA of advanced NSCLC patients | 6 months
  Analyze the driver gene mutation frequency in ctDNA from advanced NSCLC patients with tumor tissue driver gene mutation
The gene mutation coincidence rate between CTCs and ctDNA | 6 months
  Comparison the gene mutation coincidence rate between CTCs and ctDNA

CONTACTS AND LOCATIONS:
Overall Officials: Yayi He, MD,PHD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haber DA, Velculescu VE. Blood-based analyses of cancer: circulating tumor cells and circulating tumor DNA. Cancer Discov. 2014 Jun;4(6):650-61. doi: 10.1158/2159-8290.CD-13-1014. Epub 2014 May 6. PMID 24801577
- [Background] Li Y, Xu H, Su S, Ye J, Chen J, Jin X, Lin Q, Zhang D, Ye C, Chen C. Clinical validation of a highly sensitive assay to detect EGFR mutations in plasma cell-free DNA from patients with advanced lung adenocarcinoma. PLoS One. 2017 Aug 22;12(8):e0183331. doi: 10.1371/journal.pone.0183331. eCollection 2017. PMID 28829813
- [Background] Krebs MG, Metcalf RL, Carter L, Brady G, Blackhall FH, Dive C. Molecular analysis of circulating tumour cells-biology and biomarkers. Nat Rev Clin Oncol. 2014 Mar;11(3):129-44. doi: 10.1038/nrclinonc.2013.253. Epub 2014 Jan 21. PMID 24445517